CLINICAL TRIAL: NCT03662594
Title: Growth of High-Quality Oxides on The Inner Surface of ECMO Circuit by Atomic Layer Deposition to Reduce Thrombus Formation
Brief Title: Growth of High-Quality Oxides on The Inner Surface of ECMO Circuit by ALD to Reduce Thrombus Formation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 201801059DINC
Record Dates: First submitted 2018-08-26; First posted 2018-09-07 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-02

CONDITIONS: Anticoagulation
Keywords: Anticoagulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ECMO tube (Other)
  Interventions: Other: ECMO

INTERVENTIONS:
Other: ECMO — In this project, the investigators will apply a new technique of atomic layer deposition (ALD) to coat biocompatible and hemocompatible ZrO2/Al2O3 nanolaminate thin films on the inner surface of ECMO tubing to suppress the device-induced coagulopathy. ALD is a thin-film deposition technique for preparing high-quality oxides with atomic-layer accuracy. It offers many benefits including accurate thickness control. These characteristic clear accounts of the high-quality hemocompatible oxide thin films on the whole surface of complex 3-D structures, such as the inner surface The newly-prepared ECMO circuit will then undergo in vitro tests and animal study to carefully examine the safety and effectiveness of improvement of hemocompatibility.

SUMMARY:
This study evaluate thermal ALD (T-ALD) and plasma-enhance ALD (PE-ALD) processes modified cardiopulmonary bypass (CPB) tubing to investigate anticoagulation properties.

DETAILED DESCRIPTION:
ECMO is a technique which is currently being used worldwide for providing life support for patients experiencing both pulmonary and cardiac failure. Though ECMO can effectively rescue life at the initial scene, being invasive, complex, resource intensive, and serious related complications developing on the following days of ECMO support have greatly restricted it use. The major causes of ECMO-related mortality and morbidity are serious coagulopathy, either bleeding (7-34%) or thrombosis (8-17%). Contact of high extracorporeal blood flow and the large artificial surfaces plays a critical role leading to the subsequent coagulopathy. Systemic heparin and heparin-bonded circuits is usually used to reduce thrombus. However, non-urgent invasive procedures should be avoided or minimized during that support and regular clinical monitoring to guide the adjustment of optimal dosage is mandatory making the clinical care intensive. Whereas the pharmacological interventions may bring the risk of critical imbalance between hemostasis and thrombosis, efforts to modify the ECMO system focusing on improvement of biocompatibility seem a fundamental way particularly regarding the extended periods of ECMO use. ZrO2 and Al2O3 are more excellent biocompatible and hemocompatible materials compared with PVC (polyvinylchloride) which is the current material of ECMO circuit. Despite the broad applications of ZrO2 and Al2O3 in artificial implants, traditional thin-film coating techniques are unable to deposit these hemocompatible oxides on the inner surface of the PVC tubing in ECMO circuit. In this subproject, the investigators will apply a new technique of atomic layer deposition (ALD) to coat biocompatible and hemocompatible ZrO2/Al2O3 nanolaminate thin films on the inner surface of ECMO tubing to suppress the device-induced coagulopathy. ALD is a thin-film deposition technique for preparing high-quality oxides with atomic-layer accuracy. It offers many benefits including accurate thickness control, excellent conformality, high uniformity, low defect density, good reproducibility, and low deposition temperature. These characteristics clearly accounts for the feasibility to deposit high-quality hemocompatible oxide thin films on the whole surface of complex 3-D structures, such as the inner surface of ECMO tubing, using the ALD technique. The newly-prepared ECMO circuit will then undergo in vitro tests and animal study to carefully examine the safety and effectiveness of improvement of hemocompatibility.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Weighing more than 50 kg

Exclusion Criteria:

* Pregnancy
* Smoking
* Chewing betel nut
* History of any blood or cancer
* Taking anticoagulants

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-03-10 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2018-04-10 (Actual)

PRIMARY OUTCOMES:
Protein content or configuration changed | Within 3 days after blood drawed
  Use ELISA to measuring the content or configuration of a protein when blood contact material, such as human serum albumin and human plasma fibrinogen etc.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

DOCUMENTS (1):
  • Study Protocol (2018-02-22): https://cdn.clinicaltrials.gov/large-docs/94/NCT03662594/Prot_000.pdf